CLINICAL TRIAL: NCT04746417
Title: Validation of the Assessment of Skeletal Maturity Using Femoral Head in Patients With Idiopathic Scoliosis and Its Clinical Implications
Brief Title: Assessment of Skeletal Maturity Using Proximal Femoral Epiphysis in Patients With Scoliosis
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Jason Pui Yin Cheung, Clinical Associate Professor, The University of Hong Kong
Other Study IDs: FVersion 1.0
Record Dates: First submitted 2021-02-02; First posted 2021-02-09 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Idiopathic Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to explore the use of proximal femoral head for the assessment of skeletal maturity in patients with idiopathic scoliosis. The aim is to validate the use of the stages of proximal femoral epiphyseal closure in assessing pubertal growth landmarks in this patient cohort. The grading system of this skeletal maturity index will be established and its reliability and reproducibility in clinical use will be examined.

DETAILED DESCRIPTION:
There are multiple skeletal maturity measures currently in use which were established with reliability in assessing growth. The advantages and shortcomings of each index was previously examined. This study aims to explore the use of proximal femoral epiphysis, which is in close proximity of the radiographic field of the spine, in assessing the growth status of patients with idiopathic scoliosis. The stages of the proximal femoral epiphyseal ossification has been established with specific definitions. The reliability and reproducibility of using these gradings will be examined by orthopaedic surgeons. Subsequently, the assessment of different pubertal growth landmarks using these gradings will be validated, and to see whether these gradings can provide indications of peak growth and growth cessation. Finally, the relationships of such growth assessment using this proximal femoral epiphysis ossification (PFEO) system and the curve progression in idiopathic scoliosis will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic scoliosis
* Open triradiate cartilage or open distal radius epiphysis without capping

Exclusion Criteria:

* Non-idiopathic scoliosis
* Patients with growth hormone deficiency or developmental delay
* Patient has not reached skeletal maturity
* Defaulted and lost to follow-up

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients presented to our tertiary scoliosis clinic with referral for specialist consultation of scoliosis - we particularly focus on scoliosis of idiopathic nature
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
PFEO stages | 8 to 18 years
  Grade 1 to Grade 6

SECONDARY OUTCOMES:
Growth parameters | 8 to 18 years
  Standing body height
Growth parameters | 8 to 18 years
  Arm span

OTHER OUTCOMES:
Curve progression | 8 to 18 years
  Coronal Cobb angle

CONTACTS AND LOCATIONS:
Locations (1):
- Duchess of Kent Children's Hospital, Hong Kong, Hong Kong